CLINICAL TRIAL: NCT05892432
Title: Randomized, Controlled Trial of Rybelsus (Semaglutide) Among Adults With Alcohol Use Disorder (AUD)
Brief Title: Clinical Trial of Rybelsus (Semaglutide) Among Adults With Alcohol Use Disorder (AUD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-0261; R21AA031146 (NIH)
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to medication assignment, as will all care providers and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in this Arm will take a medically inert placebo. To ensure pill equivalence between groups, tablets will be packaged in the same capsule; thus, each participant will take one capsule per day. Participants will be instructed to ingest the capsule orally each morning.
  Interventions: Drug: Placebo
- Semaglutide 3 milligrams and 7 milligrams (Active Comparator): Participants in this Arm will study medication for a total of 8 weeks - on semaglutide 3 milligrams per day for 4 weeks, then 7 milligrams per day for 4 weeks. To ensure pill equivalence between groups, tablets will be packaged in the same capsule; thus, each participant will take one capsule per day. Participants will be instructed to ingest the capsule orally each morning.
  Interventions: Drug: Semaglutide 3 MG [Rybelsus]; Drug: Semaglutide 7 MG [Rybelsus]

INTERVENTIONS:
Drug: Semaglutide 3 MG [Rybelsus] — Semaglutide 3 mg will be taken for the first 4 weeks of the 8-week trial.
  Other Names: Rybelsus 3 mg
  Arms: Semaglutide 3 milligrams and 7 milligrams
Drug: Semaglutide 7 MG [Rybelsus] — Semaglutide 7 mg will be taken for the second 4 weeks of the 8-week trial.
  Other Names: Rybelsus 7 mg
  Arms: Semaglutide 3 milligrams and 7 milligrams
Drug: Placebo — A medically inert placebo medication will be taken for 8 weeks.
  Arms: Placebo

SUMMARY:
This study is a randomized controlled trial of oral semaglutide among treatment-seeking individuals with AUD. The investigators will randomly assign 50 participants to receive semaglutide (titrated to 7 milligrams (mg) per day) or matched placebo for 8 weeks. The primary aims are to assess the safety and tolerability of semaglutide in this population and to evaluate its effects, relative to placebo, on alcohol cue-elicited craving and alcohol consumption.

DETAILED DESCRIPTION:
A screening visit will be conducted at which written informed consent will be obtained and inclusion/exclusion criteria will be assessed. Subsequently, eligible participants will be randomly assigned to take oral semaglutide or matched placebo for 8 weeks, with the semaglutide dose titrated from 3 milligrams (mg)/day for the first 4 weeks to 7 milligrams (mg)/day for the second 4 weeks. Participants will complete 7 additional clinic visits (weekly during the first 4 weeks of the treatment period and biweekly during the second 4 weeks). At each visit, participants will also engage in a computerized behavioral intervention. At screening and again at the Week 6 visit, participants will complete an alcohol cue reactivity task. At the Week 1 visit, before ingesting the first dose of study medication, and again at the Week 8 visit, participants will complete a functional MRI session.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 or older.
2. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for current AUD of at least moderate severity, as assessed by the Mini International Neuropsychiatric Interview (MINI).
3. Seeking pharmacological treatment for AUD and wants to stop or cut down on drinking.
4. Has a body mass index (BMI) of at least 25 kg/m2.
5. Able to read and understand questionnaires and informed consent.
6. Lives within 50 miles of the study site.

Please contact clinical site for additional inclusion criteria.

Exclusion Criteria:

1. Current DSM-5 diagnosis of any other substance use disorder of moderate or greater severity, except for Nicotine Use Disorder, as assessed by MINI.
2. Urine drug screen at screening positive for any substance except cannabis.
3. Current DSM-5 bipolar disorder, major depressive episode, or panic disorder, as assessed by MINI.
4. Current or lifetime eating disorder (anorexia, bulimia, or binge eating disorder) or psychotic disorder, as assessed by MINI.
5. Current suicidal ideation or homicidal ideation.
6. Current use of other psychotropic medications except antidepressants (for which dose must be stable for at least the past 2 months).
7. Current or past-month use of AUD pharmacotherapy, including (e.g., oral naltrexone, acamprosate, or disulfiram) or current or past 60-day use of injectable naltrexone.
8. Current psychotherapy in which the primary focus is AUD. Attendance at Alcoholics Anonymous (AA) meetings is not exclusionary.
9. Current or past-month use of weight control medications.
10. Current or past-month use of metformin for any indication.
11. Any prior use of semaglutide or other GLP-1 agonists.
12. History of severe alcohol withdrawal (e.g., seizure, delirium tremens), as evidenced by self- report and assessment with Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar).
13. Current or lifetime Type 1 or Type 2 diabetes diagnosis, or HbA1c >6.5%.
14. Current or lifetime kidney disease or creatinine clearance <80 mL/min for participants <=55 years of age (<65 mL/min for those >55).
15. Personal history of gastrointestinal disease (e.g., gastroparesis) or pancreatitis.
16. Personal or family history of medullary thyroid carcinoma and/or multiple endocrine neoplasia syndrome type 2
17. Current or past hepatocellular disease, as indicated by verbal report or elevations of serum amylase, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of the normal range at screening.
18. Uncontrolled hypertension (systolic BP >160 mmHg or diastolic >100 mmHg).
19. Biological females of childbearing potential who are pregnant (by plasma HCG), nursing, or who are not using a reliable form of contraception.
20. Lack of a stable living situation.
21. (If participating in MRI sessions) Contraindications to MRI scanning, ferrous metal in the body including intracranial, intraorbital, or intraspinal metal, pacemakers, cochlear implants, other non-MRI-compatible devices, or other devices that could compromise the quality of the MRI images such as a permanent top retainer or braces.
22. (If participating in MRI sessions) Severe claustrophobia or morbid obesity that preclude placement in the MRI scanner.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Cue Craving Visual Analog Score | 7 weeks - change between screening and Week 6 visit
  The primary efficacy endpoint will be the magnitude of change between screening and Week 6 in the cue-craving VAS score on the first VAS item ("How strong is your craving to drink alcohol?") administered after the alcohol cue presentation. Scores range from 0 (none) to 20 (extremely strong). Higher scores indicate a higher level of craving.

SECONDARY OUTCOMES:
Number of drinks per day | 4 weeks
  The number of standard alcoholic drinks participants consume per day during the last 4 weeks of the treatment period (Week 5-8), as reported on the Timeline Follow-Back Interview.
Percentage of heavy drinking days | 4 weeks
  The percentage of heavy drinking days during the last 4 weeks of the treatment period (Week 5-8), as reported on the Timeline Follow-Back Interview.
Change in alcohol cue-elicited brain activation | 8 weeks
  Change in fMRI BOLD activation to alcohol vs. neutral beverage visual cues between baseline and Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Schacht, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual-level phenotypic data will be submitted to the NIAAA Data Archive (NDA) portal once it is available. Informed consent that allows for broad sharing of each subject's de-identified data will be obtained and personally identifiable information that allows the creation of an NDA Global Unique Identifier will be collected. The PI and study staff will work with NDA staff to specify and/or define measures to be collected, and data will be submitted in accordance with NDA submission due dates.
Time Frame: Data will become available 2 years after the grant end date, and will be available as long as the NDA exists.
Access Criteria: Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NDA data by submitting a data access request in accordance with applicable NDA policies. Data requests will be reviewed and granted by a NIAAA Data Access Committee.
URL: https://nda.nih.gov/nda/about-sharing-regimen